CLINICAL TRIAL: NCT05919680
Title: A Phase 2a, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Orziloben (NST-6179) in Subjects With Intestinal Failure-Associated Liver Disease (IFALD)
Brief Title: A Study of NST-6179 in Subjects With Intestinal Failure-Associated Liver Disease (IFALD).
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NorthSea Therapeutics B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: NST-6179-02
Record Dates: First submitted 2023-03-16; First posted 2023-06-26 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Intestinal Failure Associated Liver Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A-800 mg NST-6179 (Experimental): up to 12 subjects
  Interventions: Drug: NST-6179 Part A
- Part A matched NST-6179 placebo (Experimental): up to 6 subjects
  Interventions: Other: Matched Placebo
- Part B- 1200mg NST-6179 (Experimental): up to 12 subjects
  Interventions: Drug: NST-6179 Part B
- Part B matched NST-6179 placebo (Experimental): up to 6 subjects
  Interventions: Other: Matched Placebo

INTERVENTIONS:
Drug: NST-6179 Part A — Once daily (QD) oral administration of 800mg (32 mL solution) of NST-6179 for 4 weeks
  Arms: Part A-800 mg NST-6179
Drug: NST-6179 Part B — Once daily (QD) oral administration of 1200mg of NST-6179 for 12 weeks
  Arms: Part B- 1200mg NST-6179
Other: Matched Placebo — Matched placebo for administration in Part A or Part B
  Arms: Part A matched NST-6179 placebo; Part B matched NST-6179 placebo

SUMMARY:
This is a phase 2a, multicenter, randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of NST-6179 in subjects with intestinal failure-associated liver disease (IFALD) receiving parenteral nutrition (PN).

The study will be conducted in 2 sequential parts. Up to 36 subjects diagnosed with IFALD will be enrolled in the study, of which up to 18 subjects will be enrolled in each of the 2 parts and randomized (2:1) to receive NST-6179 (N=12/part) or matched placebo (N=6/part). Subjects in Part A will receive once daily (QD) oral administration of 800 mg (32 mL solution) NST-6179 or placebo for 4 weeks. The NST-6179 dose for Part B is planned to be 1200 mg QD for 12 weeks. Actual dose, however, will be determined during the safety review meeting.

ELIGIBILITY:
Key Inclusion Criteria:

* Adult persons aged 16 years or older at the time of informed consent.
* Minimum of 6 months on Parenteral supplementation.
* Established clinical diagnosis of IFALD based on a persistent elevation of

  1. liver enzymes (ALP, AST, ALT, or GGT ≥1.5 × upper limit of normal [ULN]) for ≥6 months and/or
  2. total bilirubin > ULN for ≥6 months.
* Laboratory parameters consistent with stable liver disease without cirrhosis as defined by:

  1. ALT and AST <5 × ULN;
  2. Total bilirubin ≤2.5 mg/dL in the absence of Gilbert's Syndrome.
  3. Serum albumin ≥2.5 g/dL;
  4. International normalized ratio (INR) ≤1.3 in the absence of anticoagulant therapy;
  5. Platelet count ≥120,000/mm3.

Key Exclusion Criteria:

* Clinical, laboratory, imaging, or histopathologic evidence of other causes of acute or chronic liver disease, including autoimmune, viral, metabolic, or alcoholic liver disease.
* Clinical evidence of compensated or decompensated hepatic cirrhosis as assessed by historical liver histology, ultrasound-based and/or signs and symptoms of hepatic decompensation (including, but not limited to, jaundice, ascites, variceal hemorrhage, and/or hepatic encephalopathy).
* Presence of hepatic impairment, end-stage liver disease, and/or a model for end-stage liver disease (MELD) score >12.
* Transient elastography read >20.0 kPA within 3 months prior to or during the Screening Period.
* Estimated glomerular filtration rate <45 mL/min based on the 2021 CKD-EPI creatinine equation.
* Poor nutritional status defined as body mass index (BMI) <17 kg/m2.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and tolerability of NST-6179 | Up to 14 Weeks
  Incidences of treatment-emergent adverse events, clinically significant chances in laboratory tests, vital signs and ECGs
To assess the pharmacokinetics of NST-6179 | Day 1 and Day 14
  area under the concentration-time curve from time 0 to last measurable concentration (AUC0-last)
To assess the pharmacodynamic effects of NST-6179 on hepatic steatosis | 12 weeks
  Relative change from baseline to week 12 in biomarkers for hepatic steatosis as measured by magnetic resonance imaging-estimated proton density fat fraction (MRI-PDFF) and controlled attenuation parameter (CAP)
To assess the pharmacodynamic effects of NST-6179 on hepatic inflammation | 12 weeks
  Absolute and relative change from baseline to week 12 in hepatic inflammation (aspartate transaminase [AST], alanine transaminase [ALT], and high sensitivity C-reactive protein [hsCRP])
To assess the pharmacodynamic effects of NST-6179 on hepatic cholestasis (bilirubin, ALP, GGT) | 12 weeks
  Absolute and relative change from baseline to week 12 in hepatic cholestasis (total bilirubin, direct bilirubin, alkaline phosphatase [ALP], and gamma-glutamyl transferase [GGT])
To assess the pharmacodynamic effects of NST-6179 on hepatic fibrosis (ELF, Pro-C3, FIB-4) | 12 weeks
  Absolute and relative change from baseline to week 12 in hepatic fibrosis as measured non-invasively by FibroScan VCTE kPa, enhanced liver fibrosis (ELF) score (and individual components), propeptide of type III collagen (PRO-C3), and fibrosis-4 (FIB-4)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Mayo Clinic Scottsdale Campus, Scottsdale, Arizona
  - University of California San Francisco Medical Center, San Francisco, California
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Emory University School of Medicine, Atlanta, Georgia
  - The University of Chicago Medical Center, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic Rochester Campus, Rochester, Minnesota
  - Mount Sinai Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - The Cleveland Clinic, Cleveland, Ohio
  - Vanderbilt University School of Medicine, Nashville, Tennessee
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No